CLINICAL TRIAL: NCT05754814
Title: SUper-Resolution Ultrasound Imaging of Erythrocytes (SURE) in Normal and Malignant Lymph Nodes
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Technical University of Denmark (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Nathalie Sarup Panduro, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: SURE-LN-2022
Record Dates: First submitted 2023-01-26; First posted 2023-03-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Cancer; Lymphoma; Lymph Node Metastasis
Keywords: head and neck cancer; lymphoma; lymph node metastasis; super-resolution ultrasound; microvasculature
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphoma; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Healthy participants
- Cases: Patients with malignant lymph nodes on the neck
  Interventions: Other: Malignant lymph nodes

INTERVENTIONS:
Other: Malignant lymph nodes — Patients with a condition; either lymphoma on the neck or head and neck cancer with lymph node metastases on the neck.
  Groups: Cases

SUMMARY:
The goal of this observational study is to visualize the small vessels in normal and cancerous lymph nodes on the neck with a new ultrasound technique.

The main questions it aims to answer are:

* Is it possible to visualize the network of the smallest vessels in lymph nodes on the neck?
* Is it possible to distinguish between healthy and cancerous lymph nodes using different parameters?

The participants will have 1-2 lymph nodes ultrasound scanned with a standard ultrasound technique and the new technique.

DETAILED DESCRIPTION:
Super-resolution ultrasound using erythrocytes (SURE) is a new ultrasound technique for visualizing the very small blood vessels in the body. The technique uses tracking of the blood's red blood cells (erythrocytes) to achieve a higher resolution of the blood vessels' shape, structure, and blood flow. The technique makes it possible to create images with much higher resolution than normal ultrasound, which means that even very small blood vessels can be imaged and measured.

In many diseases, the small blood vessels change their function or structure. One of the major disease groups where SURE has significant potential is cancer. In cancerous nodes, the small blood vessels change: they become twisted, irregular, and function poorly. If changes in the small vessels can be detected at an early stage using SURE, it can lead to quicker diagnoses and better evaluations of the effectiveness of treatment.

In this study, the investigators aim to demonstrate the practical feasibility of SURE imaging in human lymph nodes and investigate the clinical relevance of SURE imaging in the diagnosis of malignant lymph nodes by comparing lymph nodes from healthy participants with lymph nodes from participants with head and neck cancer metastases or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 70 years of age, at the time of signing the informed consent
* Participants who can lie still for 1 minute
* Capable of giving signed informed consent

Inclusion criteria for healthy participants:

* Participants who are overtly healthy as determined by medical history
* Participants who have a superficial lymph node laterally on the neck with a normal appearance on standard B-mode ultrasound available for SURE imaging

Inclusion criteria for participants with head and neck cancer or lymphoma:

* Participants who, besides their untreated head and neck cancer or lymphoma, are overtly healthy as determined by medical evaluation and medical history
* Participants with untreated lymphoma or head and neck cancer and lymph node metastasis verified by a biopsy.
* Participants who have superficial lymph nodes laterally on the neck up to 2.5 cm (so the entire lymph node is in the SURE image)
* Participants who will have their lymph nodes surgically removed

Exclusion Criteria:

* Pregnancy
* Dementia
* Physique making ultrasound scanning difficult
* Ongoing or recent (within the last 4 weeks) infectious disease (bacterial, viral, fungal, or protozoal) which may give rise to reactive lymph nodes
* Diseases that cause lymphadenopathy: Some chronic infectious diseases (HIV, Tuberculosis, Hepatitis B), Systemic diseases (rheumatoid arthritis, systemic lupus erythematosus, sarcoidosis, other rare systemic diseases*), Primary adrenal insufficiency (Addison´s disease), Leukemia, Lymphoma or other cancers (besides the type of cancer the participant is being examined for at the Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Rigshospitalet)
* Drugs that cause lymphadenopathy: Antibiotics (Cephalosporins, Penicillin, Sulfonamides), Antiepileptics (Carbamazepine, Ethosuximide, Lamotrigine, Phenytoin, Primidone), Antihypertensives (Atenolol, Captopril, Hydralazine), Other (Allopurinol, Imatinib)

  * Castleman's disease, Kikuchi's disease, Kawasaki disease, Inflammatory pseudotumor, Amyloidosis, Kimura disease, Rosai-Dorfman disease, IgG4-related disease, Still's disease, dermatomyositis, Churg-Strauss, histiocytosis, chronic granulomatous diseases, Autoimmune lymphoproliferative syndrome, lipid storage diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The healthy participants are recruited via forsøgsperson.dk and www.sundhed.dk/borger/behandling-ogrettigheder/bliv-forsoegsperson as well as via advertising posters at Rigshospitalet and at the Technical University of Denmark and possibly on social media.
  The participants will be recruited among the patients with head and neck cancer metastases or lymphoma currently referred for a fast-track program at the Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Rigshospitalet.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Super-resolution ultrasound image of normal and malignant human lymph nodes | 1 minute
  With super-resolution ultrasound imaging, the investigators will visualize the microvasculature in the lymph nodes.

SECONDARY OUTCOMES:
Vessel distribution | 1 minute
  Visual distribution of the nodal microvasculature
Microvessel density | 1 minute
  The ratio of the vessel volume to the full volume in different regions
Flow velocity | 1 minute
  In mm/s

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Sarup Panduro, MD, Principal Investigator — The Department of Diagnostic Radiology, Rigshospitalet
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen, Capital Region
  - Technical University of Denmark, Kongens Lyngby, Capital Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdeyrim A, He S, Zhang Y, Mamtali G, Asla A, Yusup M, Liu J. Prognostic value of lymph node ratio in laryngeal and hypopharyngeal squamous cell carcinoma: a systematic review and meta-analysis. J Otolaryngol Head Neck Surg. 2020 May 29;49(1):31. doi: 10.1186/s40463-020-00421-w. PMID 32471483
- [Background] Ahuja AT, Ying M, Ho SS, Metreweli C. Distribution of intranodal vessels in differentiating benign from metastatic neck nodes. Clin Radiol. 2001 Mar;56(3):197-201. doi: 10.1053/crad.2000.0574. PMID 11247696
- [Background] Andersen SB, Taghavi I, Hoyos CAV, Sogaard SB, Gran F, Lonn L, Hansen KL, Jensen JA, Nielsen MB, Sorensen CM. Super-Resolution Imaging with Ultrasound for Visualization of the Renal Microvasculature in Rats Before and After Renal Ischemia: A Pilot Study. Diagnostics (Basel). 2020 Oct 22;10(11):862. doi: 10.3390/diagnostics10110862. PMID 33105888
- [Background] Aykan NF, Ozatli T. Objective response rate assessment in oncology: Current situation and future expectations. World J Clin Oncol. 2020 Feb 24;11(2):53-73. doi: 10.5306/wjco.v11.i2.53. PMID 32133275
- [Background] Basile DP, Donohoe D, Roethe K, Osborn JL. Renal ischemic injury results in permanent damage to peritubular capillaries and influences long-term function. Am J Physiol Renal Physiol. 2001 Nov;281(5):F887-99. doi: 10.1152/ajprenal.2001.281.5.F887. PMID 11592947
- [Background] Beckman JA, Duncan MS, Damrauer SM, Wells QS, Barnett JV, Wasserman DH, Bedimo RJ, Butt AA, Marconi VC, Sico JJ, Tindle HA, Bonaca MP, Aday AW, Freiberg MS. Microvascular Disease, Peripheral Artery Disease, and Amputation. Circulation. 2019 Aug 6;140(6):449-458. doi: 10.1161/CIRCULATIONAHA.119.040672. Epub 2019 Jul 8. PMID 31280589
- [Background] Brown M, Assen FP, Leithner A, Abe J, Schachner H, Asfour G, Bago-Horvath Z, Stein JV, Uhrin P, Sixt M, Kerjaschki D. Lymph node blood vessels provide exit routes for metastatic tumor cell dissemination in mice. Science. 2018 Mar 23;359(6382):1408-1411. doi: 10.1126/science.aal3662. PMID 29567714
- [Background] Chen Q, Yu J, Rush BM, Stocker SD, Tan RJ, Kim K. Ultrasound super-resolution imaging provides a noninvasive assessment of renal microvasculature changes during mouse acute kidney injury. Kidney Int. 2020 Aug;98(2):355-365. doi: 10.1016/j.kint.2020.02.011. Epub 2020 Mar 3. PMID 32600826
- [Background] Christensen-Jeffries K, Browning RJ, Tang MX, Dunsby C, Eckersley RJ. In vivo acoustic super-resolution and super-resolved velocity mapping using microbubbles. IEEE Trans Med Imaging. 2015 Feb;34(2):433-40. doi: 10.1109/TMI.2014.2359650. Epub 2014 Sep 23. PMID 25265604
- [Background] Christensen-Jeffries K, Couture O, Dayton PA, Eldar YC, Hynynen K, Kiessling F, O'Reilly M, Pinton GF, Schmitz G, Tang MX, Tanter M, van Sloun RJG. Super-resolution Ultrasound Imaging. Ultrasound Med Biol. 2020 Apr;46(4):865-891. doi: 10.1016/j.ultrasmedbio.2019.11.013. Epub 2020 Jan 21. PMID 31973952
- [Background] Corliss BA, Mathews C, Doty R, Rohde G, Peirce SM. Methods to label, image, and analyze the complex structural architectures of microvascular networks. Microcirculation. 2019 Jul;26(5):e12520. doi: 10.1111/micc.12520. Epub 2019 Jan 17. PMID 30548558
- [Background] Demene C, Robin J, Dizeux A, Heiles B, Pernot M, Tanter M, Perren F. Transcranial ultrafast ultrasound localization microscopy of brain vasculature in patients. Nat Biomed Eng. 2021 Mar;5(3):219-228. doi: 10.1038/s41551-021-00697-x. Epub 2021 Mar 15. PMID 33723412
- [Background] Demidov V, Maeda A, Sugita M, Madge V, Sadanand S, Flueraru C, Vitkin IA. Preclinical longitudinal imaging of tumor microvascular radiobiological response with functional optical coherence tomography. Sci Rep. 2018 Jan 8;8(1):38. doi: 10.1038/s41598-017-18635-w. PMID 29311686
- [Background] Dencks S, Piepenbrock M, Opacic T, Krauspe B, Stickeler E, Kiessling F, Schmitz G. Clinical Pilot Application of Super-Resolution US Imaging in Breast Cancer. IEEE Trans Ultrason Ferroelectr Freq Control. 2019 Mar;66(3):517-526. doi: 10.1109/TUFFC.2018.2872067. Epub 2018 Sep 24. PMID 30273150
- [Background] Ehling J, Theek B, Gremse F, Baetke S, Mockel D, Maynard J, Ricketts SA, Grull H, Neeman M, Knuechel R, Lederle W, Kiessling F, Lammers T. Micro-CT imaging of tumor angiogenesis: quantitative measures describing micromorphology and vascularization. Am J Pathol. 2014 Feb;184(2):431-41. doi: 10.1016/j.ajpath.2013.10.014. Epub 2013 Nov 18. PMID 24262753
- [Background] Ehling J, Babickova J, Gremse F, Klinkhammer BM, Baetke S, Knuechel R, Kiessling F, Floege J, Lammers T, Boor P. Quantitative Micro-Computed Tomography Imaging of Vascular Dysfunction in Progressive Kidney Diseases. J Am Soc Nephrol. 2016 Feb;27(2):520-32. doi: 10.1681/ASN.2015020204. Epub 2015 Jul 20. PMID 26195818
- [Background] Errico C, Pierre J, Pezet S, Desailly Y, Lenkei Z, Couture O, Tanter M. Ultrafast ultrasound localization microscopy for deep super-resolution vascular imaging. Nature. 2015 Nov 26;527(7579):499-502. doi: 10.1038/nature16066. PMID 26607546
- [Background] Eshraghi Samani R, Shirkhoda M, Hadji M, Beheshtifard F, Hamedani SMMG, Momen A, Mollashahi M, Zendehdel K. The prognostic value of lymph node ratio in survival of head-and-neck squamous cell carcinoma. J Res Med Sci. 2018 Apr 26;23:35. doi: 10.4103/jrms.JRMS_948_17. eCollection 2018. PMID 29887903
- [Background] Foiret J, Zhang H, Ilovitsh T, Mahakian L, Tam S, Ferrara KW. Ultrasound localization microscopy to image and assess microvasculature in a rat kidney. Sci Rep. 2017 Oct 20;7(1):13662. doi: 10.1038/s41598-017-13676-7. PMID 29057881
- [Background] Harput S, Christensen-Jeffries K, Brown J, Li Y, Williams KJ, Davies AH, Eckersley RJ, Dunsby C, Tang MX, Christensen-Jeffries K, Li Y, Williams KJ, Eckersley RJ, Harput S, Dunsby C, Davies AH, Brown J, Tang MX. Two-Stage Motion Correction for Super-Resolution Ultrasound Imaging in Human Lower Limb. IEEE Trans Ultrason Ferroelectr Freq Control. 2018 May;65(5):803-814. doi: 10.1109/TUFFC.2018.2824846. PMID 29733283
- [Background] Huang C, Zhang W, Gong P, Lok UW, Tang S, Yin T, Zhang X, Zhu L, Sang M, Song P, Zheng R, Chen S. Super-resolution ultrasound localization microscopy based on a high frame-rate clinical ultrasound scanner: an in-human feasibility study. Phys Med Biol. 2021 Apr 8;66(8):10.1088/1361-6560/abef45. doi: 10.1088/1361-6560/abef45. PMID 33725687
- [Background] Jafarnejad M, Ismail AZ, Duarte D, Vyas C, Ghahramani A, Zawieja DC, Lo Celso C, Poologasundarampillai G, Moore JE Jr. Quantification of the Whole Lymph Node Vasculature Based on Tomography of the Vessel Corrosion Casts. Sci Rep. 2019 Sep 16;9(1):13380. doi: 10.1038/s41598-019-49055-7. PMID 31527597
- [Background] Jeong HS, Jones D, Liao S, Wattson DA, Cui CH, Duda DG, Willett CG, Jain RK, Padera TP. Investigation of the Lack of Angiogenesis in the Formation of Lymph Node Metastases. J Natl Cancer Inst. 2015 Jun 10;107(9):djv155. doi: 10.1093/jnci/djv155. Print 2015 Sep. PMID 26063793
- [Background] Jonasson H, Bergstrand S, Fredriksson I, Larsson M, Ostgren CJ, Stromberg T. Normative data and the influence of age and sex on microcirculatory function in a middle-aged cohort: results from the SCAPIS study. Am J Physiol Heart Circ Physiol. 2020 Apr 1;318(4):H908-H915. doi: 10.1152/ajpheart.00668.2019. Epub 2020 Mar 6. PMID 32142355
- [Background] Kierski TM, Espindola D, Newsome IG, Cherin E, Yin J, Foster FS, Demore CEM, Pinton GF, Dayton PA. Superharmonic Ultrasound for Motion-Independent Localization Microscopy: Applications to Microvascular Imaging From Low to High Flow Rates. IEEE Trans Ultrason Ferroelectr Freq Control. 2020 May;67(5):957-967. doi: 10.1109/TUFFC.2020.2965767. Epub 2020 Jan 10. PMID 31940529
- [Background] Kim E, Park JS, Son KR, Kim JH, Jeon SJ, Na DG. Preoperative diagnosis of cervical metastatic lymph nodes in papillary thyroid carcinoma: comparison of ultrasound, computed tomography, and combined ultrasound with computed tomography. Thyroid. 2008 Apr;18(4):411-8. doi: 10.1089/thy.2007.0269. PMID 18358074
- [Background] Kupferman ME, Patterson DM, Mandel SJ, LiVolsi V, Weber RS. Safety of modified radical neck dissection for differentiated thyroid carcinoma. Laryngoscope. 2004 Mar;114(3):403-6. doi: 10.1097/00005537-200403000-00002. PMID 15091209
- [Background] Lee S, Lee JY, Yoon RG, Kim JH, Hong HS. The Value of Microvascular Imaging for Triaging Indeterminate Cervical Lymph Nodes in Patients with Papillary Thyroid Carcinoma. Cancers (Basel). 2020 Oct 1;12(10):2839. doi: 10.3390/cancers12102839. PMID 33019664
- [Background] Lin F, Shelton SE, Espindola D, Rojas JD, Pinton G, Dayton PA. 3-D Ultrasound Localization Microscopy for Identifying Microvascular Morphology Features of Tumor Angiogenesis at a Resolution Beyond the Diffraction Limit of Conventional Ultrasound. Theranostics. 2017 Jan 1;7(1):196-204. doi: 10.7150/thno.16899. eCollection 2017. PMID 28042327
- [Background] Lowerison M, Zhang W, Chen X, Fan T, Song P. Characterization of Anti-Angiogenic Chemo-Sensitization via Longitudinal Ultrasound Localization Microscopy in Colorectal Carcinoma Tumor Xenografts. IEEE Trans Biomed Eng. 2022 Apr;69(4):1449-1460. doi: 10.1109/TBME.2021.3119280. Epub 2022 Mar 18. PMID 34633926
- [Background] Lowerison MR, Huang C, Lucien F, Chen S, Song P. Ultrasound localization microscopy of renal tumor xenografts in chicken embryo is correlated to hypoxia. Sci Rep. 2020 Feb 12;10(1):2478. doi: 10.1038/s41598-020-59338-z. PMID 32051485
- [Background] Maric-Bilkan C, Flynn ER, Chade AR. Microvascular disease precedes the decline in renal function in the streptozotocin-induced diabetic rat. Am J Physiol Renal Physiol. 2012 Feb 1;302(3):F308-15. doi: 10.1152/ajprenal.00421.2011. Epub 2011 Oct 26. PMID 22031855
- [Background] Opacic T, Dencks S, Theek B, Piepenbrock M, Ackermann D, Rix A, Lammers T, Stickeler E, Delorme S, Schmitz G, Kiessling F. Motion model ultrasound localization microscopy for preclinical and clinical multiparametric tumor characterization. Nat Commun. 2018 Apr 18;9(1):1527. doi: 10.1038/s41467-018-03973-8. PMID 29670096
- [Background] Pereira ER, Kedrin D, Seano G, Gautier O, Meijer EFJ, Jones D, Chin SM, Kitahara S, Bouta EM, Chang J, Beech E, Jeong HS, Carroll MC, Taghian AG, Padera TP. Lymph node metastases can invade local blood vessels, exit the node, and colonize distant organs in mice. Science. 2018 Mar 23;359(6382):1403-1407. doi: 10.1126/science.aal3622. Epub 2018 Mar 22. PMID 29567713
- [Background] Yu J, Lavery L, Kim K. Super-resolution ultrasound imaging method for microvasculature in vivo with a high temporal accuracy. Sci Rep. 2018 Sep 17;8(1):13918. doi: 10.1038/s41598-018-32235-2. PMID 30224779
- [Background] Zhu AQ, Li XL, An LW, Guo LH, Fu HJ, Sun LP, Xu HX. Predicting Axillary Lymph Node Metastasis in Patients With Breast Invasive Ductal Carcinoma With Negative Axillary Ultrasound Results Using Conventional Ultrasound and Contrast-Enhanced Ultrasound. J Ultrasound Med. 2020 Oct;39(10):2059-2070. doi: 10.1002/jum.15314. Epub 2020 May 5. PMID 32367518